CLINICAL TRIAL: NCT03987516
Title: Effects of an Active Program in Patients With Chronic Neck Pain: a Randomized Controlled Trial.
Brief Title: Active Intervention for Patients With Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0081UG
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): Patients will be included in an active intervention.
  Interventions: Other: Active exercising
- Control group (No Intervention): Patients in the control group will not receive any intervention

INTERVENTIONS:
Other: Active exercising — Patients allocated to the experimental group were included in an active exercising program adapted to each patient
  Arms: Active intervention

SUMMARY:
Neck pain is a complex biopsychosocial disorder often precipitated or aggravated by neck movements or sustained neck postures. More than 80 % of individuals experience neck pain and neck associated disorders. The aim of this study was to investigate the effects of a 4-week active exercising program in patients with chronic neck pain.

DETAILED DESCRIPTION:
While neck pain can be severely disabling and costly, treatment options have shown moderate evidence of effectiveness. The optimal physiotherapy intervention is currently unclear. Consequently, more research in this area combining different techniques in patients with a specific clinical profile is needed. It has been previously shown that participants prefer self-care measures for the management of neck pain. The aim of this study was to investigate the effects of a 4-week active exercising program in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* To suffer from chronic neck pain (at least 3 months' duration)
* Neck pain of at least 3 on a visual analogue scale.
* Participants' symptoms should be at least partly related to increased nerve mechanosensitivity in the neck and upper limb confirmed by the reproduction of participants' symptoms by median nerve upper-limb neurodynamic test.

Exclusion Criteria:

* Whiplash related neck pain.
* Previous cervical surgical intervention.
* Cognitive impairments which prevent them to follow instructions.
* Visual or acoustic limitations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-08-11 (Actual); Study Completion 2019-09-11 (Estimated)

PRIMARY OUTCOMES:
Changes in number of active trigger points | Changes from baseline to 4 weeks in the number of active trigger points assessed by palpation. The percentage of active trigger points is obtained.
  Baseline, 4 weeks

SECONDARY OUTCOMES:
Severity of pain | Changes from baseline to 4 weeks in the severity of pain assessed using the Brief Pain Inventory. The severity and the interference of pain with daily life subscales were included. Score is the sum of the items divided by the number of items.
  Baseline, 4 weeks
Functionality | Changes from baseline to 4 weeks on functionality assessed using the Neck Outcome Score.Symptoms, sleep disturbance, every day activity and pain and participation in everyday life subscales were included. They Ranged from 0 to 100 (no simptoms).
  Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Granada, Spain